CLINICAL TRIAL: NCT03678064
Title: Use of the LOK® Robotic Gait Trainer in the Early Rehabilitation of Children After an Acquired Brain Injury (ABI): A Feasibility Study - Part III
Brief Title: Use of the LOK® Robotic Gait Trainer in the Early Rehabilitation of Children After an Acquired Brain Injury (ABI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-771
Record Dates: First submitted 2018-05-03; First posted 2018-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Injury, Brain
Keywords: physical therapy; gait; pediatric rehabilitation; gross motor function; participation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lokomat (Experimental): 16 sessions total. Provided by study PT twice weekly for 8 weeks.
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — 16 sessions total. Provided by study PT twice weekly for a period of 8 weeks

SUMMARY:
After an acquired brain injury (ABI), children often require extensive physiotherapy (PT) to help them relearn to walk. There is promising evidence in pediatric neuro-motor conditions of the possibility for brain activation pattern changes in response to repetitive, task-oriented functional gait training. Robotic-assisted gait training devices such as the Lokomat (LOK) allow this type of intensive walking retraining. The aim of this study is to assess the safety, feasibility and outcome possibilities linked to a LOK intervention given as 2 of the child's 4 PT weekly sessions over 8-weeks in the early stages of rehabilitation after an ABI.

DETAILED DESCRIPTION:
This is Phase 3 of our three- year ABI Lokomat study . Phase 1 was conducted in 2016-2017 and was a single-group pre- and post-test feasibility study of the Lokomat in pediatric ABI inpatients and daypatients in which we enrolled 9 patient participants. The co-primary outcome measures for this first phase were the Gross Motor Function Measure (GMFM), Canadian Occupational Performance Measure (COPM) . Other measures of function (PEDI-CAT), gait (6 minute walk test and Timed up and GO) and individualized goals (Goal Attainment Scaling) were included. Study feasibility was evaluated via indicators such as enrollment, number of sessions completed, drop out rate, and adverse events. Phase 2 was conducted in 2017-2018 using the same core outcome set, and added a qualitative study component with child and parent and physiotherapist interviews for their perspective on the Lokomat experience and associated outcomes. The investigators enrolled 6 patient participants (quantitative and qualitative) and their caregivers (qualitative). Phase 3 will aim to enroll 6 to 8 more children to strengthen effect size estimates for the GMFM and COPM in particular (proposed co-primary outcome measures for future randomized controlled trial). The investigators will also add in a 10 metre fast walk test to allow children with lower walking tolerance to have a gait measure, and pilot a measure of children's self-efficacy that the investigators will design for this study. Finally, the investigators will take a close look at motor learning strategies (MLS) used by the PTs in both LOK and PT sessions using the validated Motor Learning Strategies Rating Instrument (MLSRI) to begin to get a profile of comparative MLS use in gym-based PT and LOK sessions. The investigators will continue to study feasibility and add to the data from the first 2 phases the ABI LOK project.

ELIGIBILITY:
Inclusion Criteria:

* Be an inpatient or daypatient in the Brain Injury Rehabilitation program at Holland Bloorview Kids Rehabilitation Hospital with moderate or severe ABI
* Be Gross Motor Function Classification System-equivalent III or IV with primary gait goals
* Have any limb distribution of involvement (spasticity or hypotonicity). The physiotherapist (PT) and Lokomat (LOK) sessions (both about 45-minutes in length) will employ a motor learning strategies approach.
* Have a femur length at least 21 cm (to fit robotic legs) and height no greater than 6' 3" to fit LOK frame
* Be no more than 12 months post-ABI (i.e., still active rehab stage), and
* Be expected by clinical team (confirmed by child's physician) to have at least 8 more weeks of inpatient or daypatient rehab
* Be able to follow Gross Motor Function Measure instructions and participate in > 45 minutes of active PT (as judged by the child's PT)
* Be able to reliably signal pain and discomfort using verbal or nonverbal signals (as assessed at the screening assessment) for LOK operation safety reasons.

Exclusion Criteria:

* A seizure in the last 12 months,
* Inability to tolerate full weightbearing
* A knee flexion contracture > 20 degrees, knee valgus >40 degrees, hip subluxation > 40% migration percentage
* Excessive tone or ataxic or dyskinetic movements may be an exclusion (would be determined at LOK set-up confirmation visit).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-66) | Baseline, 8 weeks
  Change from baseline in motor function on Gross Motor Function Measure (GMFM-66) at week 8
Canadian Occupational Performance Measure (COPM) | Baseline, 8 weeks
  Change from baseline in targeted goal abilities and satisfaction with performance as measured by the Canadian Occupational Performance Measure at week 8

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) | Baseline, 8 weeks
  Change from baseline in targeted goal abilities as measured by Goal Attainment Scaling (GAS) at week 8. Three to five individualized walking-based activity/participation goals are set with child/parent/treating PT at baseline. Goal achievement level (score of -2 to+2) evaluated by treating PT with child/parent input at post-intervention assessment. GAS outcome (achievement) is measured by a standardized T-score that is a summary score(calculated from individual goal -2 to +2 scores) for the child's set of goals . Goal accomplishment at the targeted level (averaged across the goal set) is reflected by a T score = 50.0 + 5 with range of scores from ~ 25 to 85.
Gait speed (10 minute fastest walk test ) | Baseline, 8 weeks
  Change from baseline in Gait Speed (10 minute fastest walk test) at week 8
The Pediatric Evaluation of Disability Inventory (PEDI-CAT) | Baseline, 8 weeks
  Change from baseline in PEDI-CAT at week 8.
Movement Ability Self-efficacy Questionnaire (MASQ) | Baseline, week 8
  Change from baseline in MASQ at week 8

OTHER OUTCOMES:
Feasibility indicator: Recruitment Rate | Monthly over 12 months through study completion
  Recruitment rate (%) as measured by: # of participants enrolled / # of participants screened and eligible
Feasibility indicator: Retention Rate | Monthly over 12 months through study completion
  Retention rate (%) as measured by: # of participants completing both baseline and follow-up assessment / total # of participants
Feasibility indicator: Protocol Adherence | Monthly over 12 months through study completion
  Protocol adherence (%) as measured by: Number of sessions completed / 16 possible sessions
Motor Learning Strategies Rating Instrument (MLSRI) | Week 2-3, Week 6-7
  Compare motor learning strategy (MLS) use in LOK and PT to explore how LOK use may affect motor skill acquisition post-ABI.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hung, MD, MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Virginia Wright, PT, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beretta E, Romei M, Molteni E, Avantaggiato P, Strazzer S. Combined robotic-aided gait training and physical therapy improve functional abilities and hip kinematics during gait in children and adolescents with acquired brain injury. Brain Inj. 2015;29(7-8):955-62. doi: 10.3109/02699052.2015.1005130. Epub 2015 Apr 27. PMID 25915458
- [Background] Levac D, Missiuna C, Wishart L, Dematteo C, Wright V. Documenting the content of physical therapy for children with acquired brain injury: development and validation of the motor learning strategy rating instrument. Phys Ther. 2011 May;91(5):689-99. doi: 10.2522/ptj.20100415. Epub 2011 Mar 17. PMID 21415229
- [Background] Kamath T, Pfeifer M, Banerjee-Guenette P, Hunter T, Ito J, Salbach NM, Wright V, Levac D. Reliability of the motor learning strategy rating instrument for children and youth with acquired brain injury. Phys Occup Ther Pediatr. 2012 Aug;32(3):288-305. doi: 10.3109/01942638.2012.672551. Epub 2012 May 11. PMID 22574628
- See also: Beretta E, Storm FA, Strazzer S, Frascarelli F, Petrarca M, Colazza A, Cordone G, Biffi E, Morganti R, Maghini C, Piccinini L, Reni G, Castelli E. Effect of Robot-Assisted Gait Training in a Large Population of Children With Motor Impairment Due to Cereb — https://pubmed.ncbi.nlm.nih.gov/31562873/